CLINICAL TRIAL: NCT03778047
Title: A Clinical Study for Evaluating Enzalutamide Pharmacokinetics and Pharmacodynamics, and Related Changes After Drug Switch in Chinese Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study Evaluating Enzalutamide Pharmacokinetics and Pharmacodynamics, and Related Changes After Drug Switch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hinova Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HC-1119-02
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enzalutamide (Experimental): 160mg
  Interventions: Drug: Enzalutamide
- HC-1119 (Experimental): To be determined
  Interventions: Drug: HC1119

INTERVENTIONS:
Drug: Enzalutamide — oral
  Arms: enzalutamide
Drug: HC1119 — oral
  Arms: HC-1119

SUMMARY:
This is a study for evaluating enzalutamide pharmacokinetics and pharmacodynamics, and related changes after drug switch in Chinese patients with metastatic castration-resistant prostate cancer. The study primary objective is to evaluate the pharmacokinetic characteristics of enzalutamide in Chinese patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participated in the study, with understanding of and will to comply with relevant study procedures and signed informed consent form;
2. Chinese male, ≥ 18 years old;
3. With histologically or cytologically confirmed prostate cancer, without neuroendocrine carcinoma or ductal adenocarcinoma;
4. With evidence of metastatic lesions (such as bone scan and CT/MRI);
5. Patients with relapsed, refractory, or progressive disease despite castration (surgery or chemical) or combined androgen deprivation therapy. (Progressive disease is defined as 1 or more of the following 3 criteria: PSA progression: A minimum of 3 rising PSA values with an interval of at least 1 week between determinations, resulting in a final value higher than 50% of the minimum, with a starting PSA value > 2 ng/ml; Soft tissue disease progression as defined by RECIST 1.1; Bone progression as defined by PCWG2 with 2 or more new lesions on bone scan);
6. Castrate levels of testosterone (< 50 ng/dl) at screening; bilateral orchiectomy or ongoing androgen deprivation therapy with effective GnRH analogues;
7. ECOG performance status ≤1;
8. Laboratory tests must meet the following criteria:

   1. Routine Blood Test: hemoglobin (Hb) ≥ 90g/L (no blood transfusions within 14 days prior to screening); absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelet Count (PLT) ≥ 80 x 109/L;
   2. Blood Biochemistry: creatinine (Cr) ≤ 2 x upper limit of normal (ULN), or Cr > 2 x ULN but the calculated CrCl ≥ 60 ml/min; bilirubin (BIL) ≤2 x ULN; alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤2.5 x ULN (or ≤ 5.0 x ULN for patients with liver metastases);
   3. Coagulation: INR < 1.5.
9. Estimated life expectancy > 6 months.

Exclusion Criteria:

1. Participated in other clinical drug trials within 1 month prior to screening, or the occurrence of toxicity caused by previous treatments that has not been relieved to ≤ Grade 2 toxicity (according to CTCAE 4.03) prior to enrollment;
2. Brain metastases;
3. Subjects are excluded if any of the following conditions are met:

   1. Other malignancies within the last 5 years (except for curatively treated non-melanoma skin cancer);
   2. History of organ transplants;
   3. Past medical history of seizures, serious CNS diseases, or unexplained coma, family history of seizures, or history of traumatic brain injury;
   4. Uncontrolled hypertension (systolic ≥ 160 mmHg or diastolic ≥ 100 mmHg) or other serious cardiovascular diseases. (Patients with a history of hypertension is eligible if his blood pressure is controlled with antihypertensives);
   5. Significant GI dysfunction which may affect the intake, transport, or absorption of drug (such as inability to swallow, chronic diarrhea, and bowel obstruction, etc.), or patients with complete gastrectomy;
   6. Other uncontrolled clinical diseases, including but not limited to: persistent or active infections.
4. Subjects are excluded if any of the following conditions regarding past or concomitant medication are met:

   1. Medications that lower the seizure threshold must be used during the trial;
   2. Treatment with 5α-reductase inhibitors (finasteride, dutasteride), estrogen, or cyproterone within 4 weeks prior to screening;
   3. Treatment with ketoconazole within 4 weeks prior to screening;
   4. Previously treated with investigational or approved medications that inhibit testosterone synthesis (such as abiraterone acetate, TAK-683, and TAK-448) or target testosterone receptors (such as SHR3680, proxalutamide, and ARN509), except for bicalutamide and flutamide.
5. Known hypersensitivity to any ingredient of the study drugs (enzalutamide and HC-1119) or similar drugs;
6. HIV seropositive;
7. History of medication or drug abuse;
8. Other conditions that subject is determined by the investigator to be unsuitable for this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Maximum drug concentration(Cmax) | From the first dose of the study drug to 12 weeks after dose
Time of maximum drug concentration(Tmax) | From the first dose of the study drug to 12 weeks after dose
Area under curve from time 0 to 24h (AUC0-24h) | From the first dose of the study drug to 12 weeks after dose

SECONDARY OUTCOMES:
Maximum drug concentration(Cmax) | From 13 weeks to 24 weeks after dose
Time of maximum drug concentration(Tmax) | From 13 weeks to 24 weeks after dose
Area under curve from time 0 to 24h (AUC0-24h) | From 13 weeks to 24 weeks after dose
Number of patients with adverse events | From the first dose of the study drug to 24 weeks after dose
  Safety measures
Percentage of patients with > 50% decrease in prostate specific antigen (PSA) | From the first dose of the study drug to 12 weeks after dose
  Percentage of patients with > 50% decrease in PSA levels from baseline at weeks1,3,5 6, 8, 10, and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Ethics Committee of Hunan Cancer Hospital, Changsha, China